CLINICAL TRIAL: NCT00970489
Title: (OPERA)Randomized Clinical Trial to Examine Whether Peri-operative Intake of n-3 Polyunsaturated Fatty Acids Will Reduce the Occurrence of Post-operative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Brief Title: Omega-3 Fatty Acids for Prevention of Post-Operative Atrial Fibrillation
Acronym: OPERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The OPERA Investigators (Unknown)
Responsible Party: Principal Investigator, Dariush Mozaffarian, MD, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IND-104364
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; fish oil
MeSH Terms: conditions — Atrial Fibrillation | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 fatty acid capsules (Experimental)
  Interventions: Drug: Omega -3 fatty acids
- Olive Oil capsule (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega -3 fatty acids — 10g dose of oral omega-3 fatty acid capsules over 3-5 days before surgery (or 8 g over 2 days before surgery), including the morning of surgery, followed by 2g/d after surgery for 10 days, or until discharge, whichever occurs first.
  Arms: Omega-3 fatty acid capsules
Drug: Placebo — Olive Oil capsules
  Arms: Olive Oil capsule

SUMMARY:
This is a large multi-center study to examine whether peri-operative intake of n-3 polyunsaturated fatty acids (PUFA) will reduce the occurrence of post-operative atrial fibrillation or flutter (AF) in patients undergoing cardiac surgery (CS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Scheduled for CS on the following day or later, including coronary artery bypass, valve surgery, any other open cardiac surgery (i.e., that includes opening of the pericardium), or any combination.
* Sinus rhythm on current ECG (sinus bradycardia, sinus tachycardia, and ectopy are acceptable).

Exclusion Criteria:

* Regular use (3 or more days/week) of fish oil within the past 4 weeks.
* Known allergy or intolerance to fish oil or corn oil.
* Currently pregnant.
* Unable to provide informed written consent.
* Current or planned cardiac transplant or LVAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Mozaffarian, MD DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Roberto Marchioli, MD, Principal Investigator — Laboratory of Clinical Epidemiology of Cardiovascular Disease Department of Clinical Pharmacology and Epidemiology Consorzio Mario Negri Sud Via Nazionale 8/A S. Maria Imbaro (Chieti), 66030 ITALY
Locations (1):
- US, Italy and Argentina, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Akintoye E, Sethi P, Harris WS, Thompson PA, Marchioli R, Tavazzi L, Latini R, Pretorius M, Brown NJ, Libby P, Mozaffarian D. Fish Oil and Perioperative Bleeding. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004584. doi: 10.1161/CIRCOUTCOMES.118.004584. PMID 30571332
- [Derived] Jackson JC, Mozaffarian D, Graves AJ, Brown NJ, Marchioli R, Kiehl AL, Ely EW. Fish Oil Supplementation Does Not Affect Cognitive Outcomes in Cardiac Surgery Patients in the Omega-3 Fatty Acids for Prevention of Post-Operative Atrial Fibrillation (OPERA) Trial. J Nutr. 2018 Mar 1;148(3):472-479. doi: 10.1093/jn/nxx002. PMID 29546292
- [Derived] Wu JH, Marchioli R, Silletta MG, Masson S, Sellke FW, Libby P, Milne GL, Brown NJ, Lombardi F, Damiano RJ Jr, Marsala J, Rinaldi M, Domenech A, Simon C, Tavazzi L, Mozaffarian D. Oxidative Stress Biomarkers and Incidence of Postoperative Atrial Fibrillation in the Omega-3 Fatty Acids for Prevention of Postoperative Atrial Fibrillation (OPERA) Trial. J Am Heart Assoc. 2015 May 20;4(5):e001886. doi: 10.1161/JAHA.115.001886. PMID 25994442
- [Derived] Wu JH, Marchioli R, Silletta MG, Macchia A, Song X, Siscovick DS, Harris WS, Masson S, Latini R, Albert C, Brown NJ, Lamarra M, Favaloro RR, Mozaffarian D. Plasma phospholipid omega-3 fatty acids and incidence of postoperative atrial fibrillation in the OPERA trial. J Am Heart Assoc. 2013 Oct 21;2(5):e000397. doi: 10.1161/JAHA.113.000397. PMID 24145742
- [Derived] Mozaffarian D, Marchioli R, Macchia A, Silletta MG, Ferrazzi P, Gardner TJ, Latini R, Libby P, Lombardi F, O'Gara PT, Page RL, Tavazzi L, Tognoni G; OPERA Investigators. Fish oil and postoperative atrial fibrillation: the Omega-3 Fatty Acids for Prevention of Post-operative Atrial Fibrillation (OPERA) randomized trial. JAMA. 2012 Nov 21;308(19):2001-11. doi: 10.1001/jama.2012.28733. PMID 23128104
- [Derived] Mozaffarian D, Marchioli R, Gardner T, Ferrazzi P, O'Gara P, Latini R, Libby P, Lombardi F, Macchia A, Page R, Santini M, Tavazzi L, Tognoni G. The omega-3 Fatty Acids for Prevention of Post-Operative Atrial Fibrillation trial--rationale and design. Am Heart J. 2011 Jul;162(1):56-63.e3. doi: 10.1016/j.ahj.2011.03.035. Epub 2011 Jun 12. PMID 21742090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,516 patients scheduled for cardiac surgery (CS) across 28 centers in the US, Italy, and Argentina, enrolled between Aug 2010 and Jun 2012. Inclusion criteria were broad; the main exclusions were regular use of fish oil or absence of sinus rhythm at enrollment. 48% of screened patients and 94% of eligible patients were enrolled.
Pre-assignment Details: Ineligible patients were most often excluded because they were not in sinus rhythm (40.5%), were on fish oil (28.9%), or were unwilling to provide informed consent (23.5%).
Groups:
- Olive Oil Capsule: Placebo : Olive Oil capsules All patients were randomized to receive n-3 Polyunsaturated fatty acids (PUFA) or matched placebo in equal numbers using computer-generated numbers, stratified by medical center.
  Treatment: Either oral n-3 PUFA (1 g capsules, each containing ~850 mg of EPA+DHA) or matching placebo (olive oil, 1 g capsules).
  Total loading dose = 8 g over 2 to 4 days pre-op, followed by 2 g/d post-op until hospital discharge or until post-op day 10, whichever sooner.
- Omega-3 Fatty Acid Capsules: Omega -3 fatty acids : 10g dose of oral omega-3 fatty acid capsules over 3-5 days before surgery (or 8 g over 2 days before surgery), including the morning of surgery, followed by 2g/d after surgery for 10 days, or until discharge, whichever occurs first.
Period: Overall Study
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules
Started | 758 | 758
Completed | 704 | 717
Not Completed | 54 | 41
Not completed — Death/Withdrew/Criteria Violation | 54 | 41

BASELINE CHARACTERISTICS:
Population: Patients scheduled for cardiac surgery across 28 centers in the US, Italy, and Argentina, enrolled between Aug 2010 and Jun 2012. Inclusion criteria were broad; the main exclusions were regular use of fish oil or absence of sinus rhythm at enrollment. Forty-eight percent of screened patients and 94% of eligible patients were enrolled.
Groups:
- Olive Oil Capsule: Placebo : Olive Oil capsules
- Total: Total of all reporting groups
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules | Total
Number analyzed (Participants) | 758 | 758 | 1516
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.4) | 63.8 (12.6) | 63.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 207 | 422
  Male | 543 | 551 | 1094

OUTCOME MEASURES:

1. Primary Outcome: Any First Post-op Atrial Fibrillation or Flutter (AF)
Description: Primary: Occurrence of post-CS AF (atrial fibrillation or flutter) of at least 30 seconds duration and confirmed by rhythm strip or 12-lead ECG. This will include definite AF and probable AF (SVT likely to be AF depending on rate and other characteristics).
Time Frame: up to 10 days post-surgery or discharge, whichever sooner
Measure: Number; unit: Participants
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules
Number analyzed (Participants) | 758 | 758
Participants | 233 | 227

2. Secondary Outcome: Post-op Af
Description: Secondary AF endpoints included post-op AF that was sustained (>1 hour), symptomatic, or treated with pharmacological or electrical cardioversion; post-op AF excluding atrial flutter; time to first post-op AF; and the number of post-op AF episodes per patient. OPERA also evaluated the total number of in-hospital days in which any post-op AF, including sustained post-op AF, was present; and the proportion of in-hospital days free of any post-op AF. All potential episodes of post-op AF and other tachyarrhythmias were reviewed and adjudicated by a centralized Events Committee of cardiac electrophysiologists. Additional endpoints included resource utilization, major adverse cardiovascular events (MACE), arterial thromboembolism, and 30-day mortality.
Time Frame: up to 10 days post-surgery or discharge, whichever sooner
Measure: Number; unit: Participants
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules
Number analyzed (Participants) | 758 | 758
Participants
  Sustained, symptomatic, or treated post-op AF | 231 | 224
  Post-op AF excluding flutter | 220 | 217

3. Secondary Outcome: Other Arrhythmias
Description: * The first 3 suspected episodes of atrial fibrillation or flutter of at least 30 sec duration following randomization were documented, including the following information:
    * Printed or digital rhythm strip and/or 12-lead ECG.
    * Recording of time of onset and time of cessation.
    * Additional documentation of temporally associated signs of symptoms, such as new or worsening chest pain, shortness of breath, or lightheadedness; drop in blood pressure requiring escalation of fluid or pressor treatment; or need for electrical or pharmacologic cardioversion.
  * The first suspected episode of each of other supraventricular or unknown narrow-complex tachycardia of at least 30 sec duration following randomization was also documented.
Time Frame: up to 10 days post-surgery or discharge, whichever sooner
Measure: Number; unit: Participants
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules
Number analyzed (Participants) | 758 | 758
Participants
  Other supraventricular tachycardia | 6 | 11
  Ventricular tachycardia or fibrillation | 9 | 5

4. Secondary Outcome: Other Endpoints
Description: 1. Number of days in the ICU, of telemetry monitoring, and of total hospital stay.
  2. Non-AF arrhythmias of at least 30 sec duration, including non-AF-SVT, ventricular tachycardia (VT), and ventricular flutter (VF), assessed and adjudicated by the Events Committee.
  3. MACE: Combined total mortality, myocardial infarction, and stroke.
  4. Bleeding, assessed by (a) chest tube output in the 24 hour period following surgery and (b) total number of packed red blood cell (RBC) transfusions from enrollment to end of treatment (hospital discharge or post-op day 10).
  5. Significant adverse events: Discontinuation of study treatment, at the discretion of the treating physicians, for suspected significant allergic reaction, severe gastrointestinal intolerance, significant bleeding, or other side effects requiring discontinuation.
  6. Thirty-day mortality assessed
  7. One-year mortality assessed
Time Frame: up to 10 days post-surgery or discharge, whichever sooner
Measure: Number; unit: Participants
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules
Number analyzed (Participants) | 758 | 758
Participants
  MACE, in-hospital | 20 | 13
  Total mortality, 30 days | 15 | 8

ADVERSE EVENTS:
Arm/Group | Olive Oil Capsule | Omega-3 Fatty Acid Capsules
Serious Adverse Events (participants affected / at risk) | 147/758 | 136/758
Other Adverse Events (participants affected / at risk) | 20/758 | 19/758
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olive Oil Capsule (N=758) | Omega-3 Fatty Acid Capsules (N=758)
Bleeding (Blood and lymphatic system disorders) | 36 (36) | 30 (32)
Bone marrow or coalgulation (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Cardiac (Cardiac disorders) | 54 (60) | 44 (50)
Constitutional symptoms (General disorders) | 9 (9) | 10 (10)
Dermatology or musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Gastrointestinal, hepatobiliary, or pancreas (Gastrointestinal disorders) | 4 (4) | 8 (8)
Infection (Immune system disorders) | 26 (27) | 16 (16)
Metabolic or laboratory (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Neurologic (Nervous system disorders) | 15 (17) | 10 (10)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 18 (18)
Renal or genitourinary (Renal and urinary disorders) | 6 (6) | 6 (6)
Vascular (Vascular disorders) | 3 (4) | 5 (5)
Other (General disorders) | 6 (6) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olive Oil Capsule (N=758) | Omega-3 Fatty Acid Capsules (N=758)
Bone marrow or coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Cardiac (Cardiac disorders) | 3 (3) | 6 (6)
Constitutional symptoms (General disorders) | 1 (1) | 0 (0)
Dermatology or musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Gastrointestinal, hepatobiliary, or pancreas (Gastrointestinal disorders) | 2 (2) | 8 (8)
Infection (Immune system disorders) | 1 (1) | 1 (1)
Metabolic or laboratory (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Neurologic (Nervous system disorders) | 5 (5) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Renal or genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Vascular (Vascular disorders) | 1 (1) | 0 (0)
Other (General disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Best-practice guidelines for preventing post-op atrial fibrillation were recommended to Centers. The duration prior to surgery may have been too short to be effective; or the dose of n-3 PUFA too low to produce benefit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No